CLINICAL TRIAL: NCT07236554
Title: Blood Flow Restriction Training Versus Mulligan Technique in Treatment of Lateral Epicondylitis : a Randomized Controlled Trial
Brief Title: Blood Flow Restriction Training Versus Mulligan Technique in Treatment of Lateral Epicondylitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nasr Awad Abdelkader Othman, Professor of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/006094
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Lateral Epicondylitis (Tennis Elbow)
MeSH Terms: conditions — Tennis Elbow | interventions — Blood Flow Restriction Therapy; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- BFRT Group (A) (Experimental): Low-load resistance training with blood flow restriction (BFR)
  Interventions: Device: blood flow restriction
- MWM Group (B) (Active Comparator): In addition to home exercises, the MWM group performed MWM
  Interventions: Other: Mulligan's with mobilization
- Control group (C) (Placebo Comparator): Stretching and strengthening exercises for the forearm extensors
  Interventions: Other: Exercise

INTERVENTIONS:
Device: blood flow restriction — The physical therapist will apply the occlusive cuff on the upper arm (brachium) with a pressure of 0.5 times of patient's systolic blood pressure. The physiotherapist will use the BFR cuffs from SAGA
  Arms: BFRT Group (A)
Other: Mulligan's with mobilization — First, the pain-free angle of application will be determined for each patient. The lateral condyle of the humerus will be fixed by the first bar space of the physiotherapist. The elbow joint will be glided until no pain will be felt in the elbow joint and the hand will be in the contracted position.
  Arms: MWM Group (B)
Other: Exercise — Eccentric training for the extensor carpi radialis brevis muscle, the most affected wrist extensor tendon, and static stretching exercises for the extensor carpi radialis brevis muscle will be provided as a home exercise program.
  Arms: Control group (C)

SUMMARY:
The purpose of this study is to evaluate the effectiveness of blood flow restriction training (BFRT) verses Mulligan's technique in improving pain, grip strength, and functional outcomes in patients with lateral epicondylitis (LE).

DETAILED DESCRIPTION:
Lateral epicondylitis (LE) is a work-related musculoskeletal disorder caused by the tendon's inflammation of either one or both of the extensor carpi radialis longus and extensor carpi radialis brevis. It is often referred to tennis elbow. It manifests as pain on the lateral side of the elbow and reduced range of motion, which results in weakening and impairment in the forearm muscles (Ahmad et al., 2013).With no sex predisposition, LE is a widespread ailment that affects up to 3% of the population (Vaquero-Picado et al., 2017). Etiological factors of LE include overuse, repetitive movements, physically forceful occupational activities, exercise errors, misalignments, flexibility problems, ageing, muscle imbalances and psychological (e.g. job strain) factors. The estimated incidence of LE ranges from 2.0-11.3 per 100 worker-years in specific activity sectors (Herquelot et al., 2013; Bongers et al., 2002).

ELIGIBILITY:
Inclusion Criteria:

1) 36 subjects of both gender aged between 18 and 50 years with a positive test of LE (Positive Cozen's, Maudsley's, and/or Mill's test), which has been determined based on physical therapy assessment procedures; 2) the presence of pain in the lateral epicondyle of the humeral bone; and 3) show decreased muscle strength and functional ability.

Exclusion Criteria:

While the exclusion criteria of this study will be 1) refusal to be a sample in this study; 2) presences of bilateral symptoms; 3) presences of sensory and motor impairment of the upper extremities; 4) samples with systemic disease and metabolic disorders; 5) history of trauma and surgery on the elbow; 6) having a history of malignancy and peripheral vascular disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Grip strength | 4 weeks
  The patients' maximal grip strength will be measured with a hand dynamometer.
Pain intensity | 4 weeks
  Measured using an 11-point numeric pain-rating scale.
Patient-Rated Tennis Elbow Evaluation (PRTEE) Score | 4 weeks
  Measures pain and disability (0-100 scale, with 100 = worst pain & disability).

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr.Nasr A Abdelkader, professor, Principal Investigator — Cairo Univesity
Locations (1):
- Faculty of Physical Therapy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT07236554/Prot_SAP_ICF_000.pdf